CLINICAL TRIAL: NCT00407589
Title: Systemic Pharmacokinetics of BOL-303224-A After Single and Multiple Instillations of BOL-303224-A in Subjects With Suspected Bacterial Conjunctivitis
Brief Title: Systemic Pharmacokinetics of BOL-303224-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 478-PK
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Conjunctivitis, Bacterial
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — besifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BOL-303224-A (Experimental): Systemic exposure of BOL-303224-A following single and multiple topical doses
  Interventions: Drug: BOL-303224-A

INTERVENTIONS:
Drug: BOL-303224-A — 1 drop in each eye, TID for 5 days at approximately 6 h intervals, with a final, single dose on the morning of Visit 7 (Day 6).
  Other Names: ISV-403; Besifloxacin

SUMMARY:
This is a multi-center, open-label, single dose/multiple dose, pharmacokinetic study in participants with bacterial conjunctivitis. The purpose of this study is to determine the extent of systemic exposure to BOL-303224-A following single and multiple topical administration of BOL-303224-A in participants with suspected bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* must be at least 18 years of age, any race
* must have a clinical diagnosis of acute bacterial conjunctivitis and exhibit purulent conjunctival discharge and redness in both eyes
* women of childbearing potential must utilize reliable contraceptive methods and have a negative pregnancy test

Exclusion Criteria:

* Pregnant or nursing women
* known hypersensitivity to fluoroquinolones or to any of the ingredients in the study medication
* use of any antibiotic within 72 hours of enrollment
* participation in an ophthalmic drug or devise research study within 30 days prior to entry in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assessment of systemic pharmacokinetics following a single dose and steady-state pharmacokinetics after multiple TID dosing | Blood samples will be collected from 0 to 6 hours on Day 1 and from 0 to 12 hours on Day 6. There will be additional sampling times at 0 hours on Day 2-5.

SECONDARY OUTCOMES:
Investigator ratings of ocular discharge and bulbar conjunctival injection, Visual Acuity, ophthalmoscopy findings and Adverse event collection | Througout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Cornerstone Eyecare, High Point, North Carolina, United States